CLINICAL TRIAL: NCT04228471
Title: Early PReserved SPONtaneous Breathing Activity in Mechanically Ventilated Patients With Acute Respiratory Distress Syndrome - The PReSPON Randomized Controlled Trial
Brief Title: Early PReserved SPONtaneous Breathing Activity in Mechanically Ventilated Patients With ARDS (PReSPON)
Acronym: PReSPON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, Christian Putensen, Principal Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKB_PReSPON
Record Dates: First submitted 2019-12-19; First posted 2020-01-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Airway Pressure Release Ventilation; Bilevel Continuous Positive Airway Pressure; Biphasic Continuous Positive Airway Pressure; Mechanical Ventilation; Ventilator-Induced Lung Injury; Spontaneous Breathing
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous Breathing Group (Experimental): Spontaneous breathing activity will be allowed during APRV within one hour after randomization throughout the first 48 hours.
  After 48 hours, standard routine care should be provided in both groups, although we suggest moderate sedation while spontaneous breathing is maintained with APRV, pressure support ventilation (PSV), or other assisting ventilator modes. Weaning off mechanical ventilation will be performed after 48 hours according to a protocol using spontaneous breathing trials.
  Interventions: Procedure: spontaneous breathing activity during APRV
- Controlled Mechanical Ventilation Group (Experimental): Pressure controlled mechanical ventilation will be applied throughout the first 48 hours.
  After 48 hours, standard routine care should be provided in both groups, although we suggest moderate sedation while spontaneous breathing is maintained with APRV, pressure support ventilation (PSV), or other assisting ventilator modes. Weaning off mechanical ventilation will be performed after 48 hours according to a protocol using spontaneous breathing trials.
  Interventions: Procedure: No spontaneous breathing activity

INTERVENTIONS:
Procedure: spontaneous breathing activity during APRV — Allowing spontaneous breathing activity with APRV throughout the first 48 hours.
  Arms: Spontaneous Breathing Group
Procedure: No spontaneous breathing activity — No spontaneous breathing activity will be allowed with pressure controlled ventilation throughout the first 48 hours.
  Arms: Controlled Mechanical Ventilation Group

SUMMARY:
The potential benefits of preserved early spontaneous breathing activity during mechanical ventilation are an increased aeration of dependent lung regions, less need for sedation, improved cardiac filling, and better matching of pulmonary ventilation and perfusion and thus oxygenation. Two small randomized controlled trials (RCTs) in patients with acute respiratory distress syndrome (ARDS) reported less time on mechanical ventilation and in the intensive care unit (ICU) with preserved early spontaneous breathing activity during Airway Pressure Release Ventilation (APRV).

Debate exists over the net effects of preserved early spontaneous breathing activity with regard to ventilator-associated lung injury (VALI). In fact, by taking advantage of the potential improvement in oxygenation and recruitment at lower inflation pressures associated with APRV, physicians could possibly reduce potentially harmful levels of inspired oxygen, tidal volume, and positive end-expiratory pressure (PEEP). However, spontaneous breathing during mechanical ventilation has the potential to generate less positive pleural pressures that may add to the alveolar stretch applied from the ventilator and contribute to the risk of VALI. This has led to an ongoing controversy whether an initial period of controlled mechanical ventilation with deep sedation and neuromuscular blockade or preserved early spontaneous breathing activity during mechanical ventilation is advantageous with respect to outcomes in ARDS patients.

A RCT investigating the effects of early spontaneous breathing activity on mortality in moderate to severe ARDS has been highly recommended in the research agenda for intensive care medicine.

The objective of this study is to evaluate the efficacy and safety of preserved spontaneous breathing activity during APRV in the early phase of moderate to severe ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe ARDS for ≤ 48 hours according to the Berlin definition will be defined by acute onset of:

   1. PaO2/FiO2 ≤ 200 mmHg (equivalent to ≤ 26.7 kPa) under invasive mechanical ventilation with PEEP ≥ 5 cmH2O
   2. Bilateral infiltrates documented by chest radiograph
   3. Not fully explained by cardiac failure or fluid overload (e.g. echocardiography)
2. Requirement for positive pressure ventilation via an endotracheal tube/ tracheotomy
3. Presence of informed consent according to local regulations
4. Age ≥ 18 years
5. Expected duration of mechanical ventilation > 48 hours at randomization

Exclusion Criteria:

1. Need of extracorporeal lung support, high frequency oscillation and/or inhaled vasodilators for severe hypoxemia prior to inclusion
2. Woman known to be pregnant, lactating or having a positive or indeterminate pregnancy test
3. Neuromuscular disease that impairs ability to ventilate spontaneously
4. Severe chronic respiratory disease (e.g. COPD, pulmonary fibrosis, and other chronic diseases of the lung, chest wall or neuromuscular system) requiring home oxygen therapy or mechanical ventilation (non-invasive ventilation or via tracheotomy) except for Continuous Positive Airway Pressure (CPAP) or non-invasive Biphasic Positive Airway Pressure (BiPAP) used solely for sleep-disordered breathing
5. Chronic kidney disease stage V (requirement of dialysis) according to the K/DOQI definition of chronic kidney disease
6. Massive diffuse alveolar haemorrhage
7. Recent lung transplant < 12 months
8. Morbid obesity defined as weight greater than 1 kg / cm
9. Burns > 70% total body surface
10. Suspected or known elevated intracranial pressure
11. Chronic liver disease (Child-Pugh grade C)
12. Ongoing chemotherapy and/or bone marrow transplantation within the last 3 months
13. Moribund patient not expected to survive 48 hours
14. Patients not expected to survive 90 days on the basis of the premorbid health status
15. Patient, surrogate, or physician not committed to full life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at study day 28 (D28) | All-cause mortality at D28 will be defined as number of patients who deceased at day 28.
  All-cause mortality at D28 will be defined as number of patients deceased at D28 divided by number of all patients. In case of missing survival status in more than 1% of the patients, additional analyses will be carried out using multiple imputation or estimating-equation methods. The date of death will be recorded for all patients who die. Up to D28, the patient's location at the time of death (ICU or hospital) will also be recorded.
Number of Ventilator Free Days (VFD) until day 28 (D28) | Number of Ventilator Free Days will be measured until day 28.
  Number of VFDs until D28 are defined as number of days alive and completely off the ventilator until day 28. A patient will be reported as ventilator free after two consecutive calendar days of unassisted spontaneous breathing (UAB).
  UAB is defined as:
  * Spontaneously breathing with face mask, nasal prong oxygen or room air
  * T-piece breathing
  * Tracheostomy breathing
  * CPAP ≤5 cmH2O without pressure support or another mode of assisted mechanical ventilation
  * Use of CPAP or BIPAP solely for sleep apnoea management
  Patients still on positive pressure ventilation/receiving assisted breathing who are transferred to another hospital or healthcare facility prior to D28 will be followed up to assess the VFD outcome at D28.

SECONDARY OUTCOMES:
All-Cause Mortality Rate at study day 90 (D90) | All-cause mortality at D90 will be defined as number of patients who deceased at day 90.
  All-cause mortality at D90 is defined as number of patients deceased at D90 divided by number of all patients. Patients with missing survival status will be counted as non-survivor.
Number of Vasoactive Drug Free Days until study day 28 (D28) | Number of Vasoactive Drug Free Days will be measured until D28.
  Number vasoactive drug free days are defined as number of days alive and completely off the vasoactive drugs until D28. Any vasoactive support given to the patient will be recorded in the e-CRF. Vasoactive support includes: catecholamine and non-catecholamine vasopressors, inotropes and vasodilating agents.
Number of Renal Support Free Days until study day 28 (D28) | Number of Renal Support Free Days will be measured until study day 28.
  Number of Renal Support Free Days are defined as number of days alive and completely off the renal support until day 28. Any renal support given to the patient will be recorded on a specific page in the e-CRF.
Sequential Organ Failure Assessment (SOFA) | The score will be assessed pre-randomization on study day 1 (D1) and daily up to study day 7 (D7) and while the patient is in the ICU until D28.
  Organ failure status will be assessed using the mean SOFA score, which assesses six organ systems: respiration, coagulation, liver, cardiovascular, central nervous system and renal function. A patient will be defined as being free of organ failure when the SOFA score is zero.

OTHER OUTCOMES:
Level of Sedation until study day 7 (D7) | For each study day, the distribution of Ramsay scale, Richmond Agitation-Sedation Scale, or Riker Sedation-Agitation Scale and the number of patients deviating from the target will be described until D7.
  Level of Sedation will be determined using the Ramsay scale [minimum value: 1 (anxious, agitated, restless) to 6 (no response to light glabellar tap or loud auditory stimulus)], the Richmond Agitation- Sedation Scale [minimum value: -5 (unarousable) to +4 (combative)], or the Riker Sedation-Agitation Scale [minimum value: 1 (unarousable) to 7 (dangerous agitation)].
  Sedation/analgesia according to local standard will be titrated to achieve either a deep or a moderate sedation level. Deep sedation is defined as a Ramsay score of 5 to 6, which corresponds to a Richmond Agitation-Sedation Scale (RASS) of -4 to -5 or a Riker Sedation-Agitation Scale of 1 to 2. Moderate sedation is defined as a Ramsay score of 2 to 3, which corresponds to a RASS of 0 to -1 or a Riker Sedation-Agitation Scale of 3 to 4.
Level of Analgesia until study day 7 (D7) | The distribution of Behavioural Pain Scale will be described for each study day until D7.
  Level of analgesia will be determined using the Behavioural Pain Scale for pain assessment in intubated patients. The Behavioral Pain Scale quantifies pain using body language and patient-ventilator interactions for intubated patients. Minimum value: 3 (calm, no pain), maximum value: 12 (maximum pain, restless).
Occurrence of barotrauma w/o Chest Tube until ICU discharge or study day 28 (D28) | The number of patients with barotrauma will be counted until ICU discharge or D28 whatever comes first.
  Barotrauma will be defined as newly developed pneumothorax, pneumomediastinum, subcutaneous emphysema, or pneumatocele larger than 2 cm in diameter with and without a chest tube and will be reported as adverse event (AE).
Occurrence of pneumonia until ICU discharge or study day (D28) | Will be counted until ICU discharge or D28 whatever comes first.
  Any newly acquired pneumonia either microbiologically confirmed or radiologically and clinically suspected by the American Thoracic Society definition requiring antimicrobial treatment.
Weaning Failure until study day 28 (D28) | Will be measured until D28.
  Weaning failure will be reported as failure to pass SBTs until D28. The proportion of patients with weaning failure will be analyzed.
Use of Prone Positioning until study day 28 (D28) | Will be counted until D28.
  Prone positioning will be recorded until study day 28 (D28). The proportion of patients with prone positioning will be analyzed.
Use of Extra-corporeal Membrane Oxygenation (ECMO) as a rescue therapy until study day 28 (D28) | Use of Extra-corporeal Membrane Oxygenation (ECMO) will be counted until study day 28 (D28).
  In refractory hypoxemia (PaO2/FIO2 < 60 mmHg) and in patients who do not respond with a substantial increase in arterial oxygenation in the transition from lower to higher PEEP a rescue therapy is allowed. The proportion of patients with Extra-corporeal Membrane Oxygenation (ECMO) will be analyzed.
Use of an inhaled vasodilator (e.g. inhaled nitric oxide) as a rescue therapy until study day 28 (D28) | Use of an inhaled vasodilator will be counted until study day 28 (D28).
  In refractory hypoxemia (PaO2/FIO2 < 60 mmHg) and in patients who do not respond with a substantial increase in arterial oxygenation in the transition from lower to higher PEEP a rescue therapy is allowed. The proportion of patients with the use of an inhaled vasodilator will be analyzed.
Use of an neuromuscular blocking agent (NMBA) (if not in the Control Group) as a rescue therapy until study day 28 (D28) | Use of an neuromuscular blocking agent (NMBA) (if not in the Control Group) will be counted until study day 28 (D28).
  In refractory hypoxemia (PaO2/FIO2 < 60 mmHg) and in patients who do not respond with a substantial increase in arterial oxygenation in the transition from lower to higher PEEP a rescue therapy is allowed. The proportion of patients with the use of an neuromuscular blocking agent (NMBA) (if not in the Control Group) will be analyzed.
Use of high-frequency oscillation as a rescue therapy until study day 28 (D28) | Use of high-frequency oscillation will be counted until study day 28 (D28).
  In refractory hypoxemia (PaO2/FIO2 < 60 mmHg) and in patients who do not respond with a substantial increase in arterial oxygenation in the transition from lower to higher PEEP a rescue therapy is allowed. The proportion of patients with the use of high-frequency oscillation will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Putensen, M.D., PhD., Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Department of Anesthesiology and Critical Care Medicine, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided